CLINICAL TRIAL: NCT05802511
Title: Post Market Study of Exablate Model 4000 Type 1.0/1.1 Following the Treatment of Neuropathic Pain
Brief Title: Study of Exablate Model 4000 Type 1.0/1.1 Following the Treatment of Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP003
Record Dates: First submitted 2023-03-15; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Neuropathy; Neuropathic Pain
MeSH Terms: conditions — Peripheral Nervous System Diseases; Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exablate treatment (Experimental): Exablate treatment on Neuropathic Pain
  Interventions: Device: Exablate treatment

INTERVENTIONS:
Device: Exablate treatment — Exablate treatment for Neuropathic Pain

SUMMARY:
The Exablate 4000 obtained CE Mark for the treatment of Neuropathic Pain in December 2012. The purpose of this post market study is to obtain real world data on the safety and performance of the Exablate treatment for neuropathic pain.

The objective of this study is to capture the change in pain intensity, physical/emotional function, and pain impact for patients diagnosed with neuropathic pain who undergo an Exablate treatment.

DETAILED DESCRIPTION:
The purpose of this post market study is to obtain real world data on the safety and performance of the Exablate treatment for neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 30 years or older
* Subject undergoing an Exablate procedure for their planned neuropathic treatment per local institution standard of care
* Subject has diagnosis of "definite" neuropathic pain (grading system IASP-NeupSIG)
* Patient has a score of 6 or higher on the Numeric Rating Scale (NRS)
* Subject has tried and failed at least three documented medically supervised treatments (including, but not limited to physical therapy, acupuncture, etc.) and has failed medication treatment from at least two different medication classes
* Subject's pain-related medication regimen is stable 4 weeks prior to the baseline evaluation
* Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all study visits

Exclusion Criteria:

* Subject diagnosed with a nociceptive chronic pain syndrome
* Subject does not agree to participate or is unlikely to participate for the entirety of the study
* Subject is currently participating in another clinical investigation with an active treatment arm

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Pain Numerical Rating Score (NRS) | 72 h
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. The subjects will be asked to rate their average pain over the past 24 hours specific to the area(s) of the pain being treated on a 0 (no pain) to 10 (worst imaginable pain) scale. A higher score indicates a higher pain level.
Pain Numerical Rating Score (NRS) | 1 month
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. The subjects will be asked to rate their average pain over the past 24 hours specific to the area(s) of the pain being treated on a 0 (no pain) to 10 (worst imaginable pain) scale. A higher score indicates a higher pain level.
Pain Numerical Rating Score (NRS) | 3 months
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. The subjects will be asked to rate their average pain over the past 24 hours specific to the area(s) of the pain being treated on a 0 (no pain) to 10 (worst imaginable pain) scale. A higher score indicates a higher pain level.
Pain Numerical Rating Score (NRS) | 12 months
  The pain NRS consists of 1 question that will be asked by interviewing the subjects. The subjects will be asked to rate their average pain over the past 24 hours specific to the area(s) of the pain being treated on a 0 (no pain) to 10 (worst imaginable pain) scale. A higher score indicates a higher pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Centro Neurolesi "Bonino-Pulejo", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided
sponsor